CLINICAL TRIAL: NCT03604432
Title: Prophylactic Limited Left Sided Maze Procedure to Prevent Post-operative Atrial Fibrillation in Adult Cardiac Surgery Patients
Brief Title: Prophylactic Maze to Prevent Atrial Fibrillation in Adult Cardiac Surgery
Acronym: PREVENT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Charles Willekes, Cardiothoracic Surgeon, Corewell Health West
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-157
Record Dates: First submitted 2018-06-19; First posted 2018-07-27 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Control group (No Intervention): Electric cardiac surgery only
- Treatment group (Experimental): Elective cardiac surgery plus prophylactic maze procedure
  Interventions: Device: propylactic maze

INTERVENTIONS:
Device: propylactic maze — Prophylactic limited left sided maze procedure for subjects in the treatment arm
  Other Names: Atricure synergy ablation system
  Arms: Treatment group

SUMMARY:
This study will look at performing a prophylactic limited left sided maze procedure during concomitant adult cardiac surgery to prevent the common occurrence of postoperative atrial fibrillation.

DETAILED DESCRIPTION:
This is a prospective, single site, randomized, small feasibility study using a FDA approved device for a new indication. Subjects undergoing a CABG, AVR, or CABG/AVR will be randomized 1 to 1 to a control or treatment group. The control group will undergo their index cardiac surgery procedure only. The treatment group will undergo their index cardiac procedure along with a limited left sided maze procedure. The maze procedure will be done with the Atricure synergy ablation system. This is an FDA approved device that will be used for this new indication.

The left sided limited maze procedure will consist of pulmonary vein isolation and removal of the left atrial appendage.

A total of 60 subjects will be enrolled in this study at a single site.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery
* AVR
* CABG
* AVR/CABG

Exclusion Criteria:

* History of AF/Aflutter
* Less common cardiac surgeries:
* aortic root replacement
* aortic dissections
* myxoma
* pericardectomies
* off-pump procedures
* redo procedures
* Subjects with existing pacemakers, AICD
* Vulnerable population
* Emergent surgery
* Currently participating in investigational drug or device study.
* Subjects currently on antiarrhythmic drugs Class I and III including amiodarone.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Willekes, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Hospitals, Grand Rapids, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Elective cardiac surgery only
- Treatment Group: Elective cardiac surgery plus prophylactic maze procedure
  prophylactic maze: Prophylactic limited left sided maze procedure for subjects in the treatment arm
Period: Overall Study
Arm/Group | Control Group | Treatment Group
Started | 31 | 29
Completed | 31 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Full Range); unit: years] | 75 [71 to 79] | 75 [71 to 79] | 75 [71 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 24 | 15 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Documented Post-operative Atrial Fibrillation
Description: Per the STS registry definition of occurrence of postoperative atrial fibrillation that requires treatment.
Time Frame: From date of index surgical procedure to date of discharge, on average 1 week.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 31 | 29
Participants | 17 | 2

2. Secondary Outcome: Number of Participants Requiring Antiarrhythmic Medications in the Treatment Group Versus Control Group
Description: the utilization of antiarrhythmic medication required to manage postoperative atrial fibrillation will be recorded
Time Frame: immediately after procedure/surgery up to discharge from the hospital, average 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 31 | 29
Participants | 14 | 2

3. Secondary Outcome: Percentage of Adverse Events Related to Use of the Radiofrequency Device or Left Atrial Appendage Amputation.
Description: record and describe any patient related morbidity or adverse outcome related to the radiofrequency pulmonary vein isolation or left atrial appendage removal
Time Frame: during the procedure/surgery, up to 8 hours
Measure: Mean (Standard Deviation); unit: percentage of events
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 31 | 29
percentage of events | 0 (0) | 0 (0)

4. Secondary Outcome: Number of Participants Requiring Anticoagulants Medications in the Treatment Group Versus Control Group
Description: the utilization of anticoagulant medications required to manage postoperative atrial fibrillation will be recorded
Time Frame: immediately after procedure/surgery up to discharge from the hospital, on average 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 31 | 29
Participants | 7 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 15/31 | 12/29
Other Adverse Events (participants affected / at risk) | 23/31 | 21/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=31) | Treatment Group (N=29)
Post op Atrial Fibrillation (Cardiac disorders) | 6 (6) | 1 (1)
Acute Kidney Injury/ Acute Renal Failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Respiratory Infections/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Covid 19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Atrial Flutter (Cardiac disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 0 (0) | 2 (2)
Thrombotic Event (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
ulcerated aorta (Vascular disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Conduit Issues (Cardiac disorders) | 0 (0) | 2 (2) — angioplasty and stent required post-op; coronary artery occlusion
PEA Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension/systemic (Cardiac disorders) | 0 (0) | 1 (1)
GI disorders (Gastrointestinal disorders) | 2 (2) | 0 (0) — colitis; ogilvie syndrome
Miscellaneous (General disorders) | 4 (5) | 1 (2) — cellulitis, deconditioning, lens discoloration, cholecystitis, leg pain, skin melanoma, osteo arthritis
injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — fall and fracture.
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
neurological disorder (Psychiatric disorders) | 2 (2) | 0 (0) — encephalopathy;delirium
Dysphagia (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute brain infarct (Vascular disorders) | 1 (1) | 0 (0)
Carotid Stenosis (Vascular disorders) | 1 (1) | 0 (0) — known pre-op but led to intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=31) | Treatment Group (N=29)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Bone Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 11 (11)
Confusion/Delerium (Nervous system disorders) | 4 (4) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Contusion (Vascular disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Post op Afib (Cardiac disorders) | 12 (12) | 0 (0)
Elevated Creatine (Renal and urinary disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT03604432/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT03604432/ICF_001.pdf